CLINICAL TRIAL: NCT01959360
Title: Minimal Invasive Surgery in Total Hip Arthroplasty Patients; Strength, Functionality and Post Operative Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100889
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Hip Osteoarthritis
Keywords: Arthroplasty, Total Hip Replacement, Hip; Surgical Procedures, Operative; Surgical Procedures, Minimally Invasive
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- direct lateral (Active Comparator)
  Interventions: Procedure: Direct lateral
- minimal invasive (Experimental)
  Interventions: Procedure: minimal invasive
- modified minimal invasive (Experimental)
  Interventions: Procedure: modified minimal invasive

INTERVENTIONS:
Procedure: Direct lateral — Total hip replacement; direct lateral approach
  Arms: direct lateral
Procedure: minimal invasive — Total hip replacement; minimal invasive approach
  Arms: minimal invasive
Procedure: modified minimal invasive — Total hip replacement; modified minimal invasive approach
  Arms: modified minimal invasive

SUMMARY:
The aim of the present study is to explore the most efficient surgical approach in total hip replacement in short and long term when concerning strength, functionality and postoperative complications.

The objective is to register muscular strength, hip joint functionality/mobilisation and complications after total hip arthroplasty (THA) performed by two minimal invasive/incision surgeries (MIS) versus the traditionally lateral approach.

The primary working hypothesis is that due to a minimal dissection and reduced trauma in the muscles, patients will tolerate early hospital discharge better after MIS than after traditional lateral surgery. Patients in the MIS group will also be more active and maintain muscular strength and hip joint functionality/mobilisation better than patients in the lateral group.

DETAILED DESCRIPTION:
With total hip replacement surgery, the orthopaedic surgeon's aim is not only pain relief for the patient, but also restoration of hip joint biomechanics resulting in a minimal functional deficit and maximal longevity of the implant. It is not exceptional that these patients still experience mild to moderate long-term impairments postoperatively. These impairments include pain, muscle weakness of the hip abductors, contracture of the hip, gait disorders, as well as weakness of hip extensors and flexors. These problems may in turn lead to complications such as joint instability and loosening of the implant. When the lateral surgical approach is used, major concerns after total hip replacement surgery are muscle abductor weakness/atrophy, tendon defects of the gluteus minimus muscle, and unsuccessful reattachment or denervation of the anterior gluteal flap.

Minimal incision/invasive surgery (MIS) is defined as a surgical approach performed through a short skin and muscle incision to avoid injury to muscles and tendons. Following minimally invasive approach reduced muscle trauma has been found. Moreover clinical outcome improved, as the gluteus medius muscle can be spared more successfully. However, it is debated whether or not the overall results of MIS are superior, or even as good as the traditional hip replacement surgery in terms of component placing and time to revision of the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for THA
* Diagnosis of primary osteoarthritis as the main cause for elective THA
* American Society of Anesthesiologists (ASA) score I, II, and stable III

Exclusion Criteria:

* Musculoskeletal diseases
* Current heart/pulmonary- or malignant diseases likely to influence the physical testing performance.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Implant stability | 2 years

SECONDARY OUTCOMES:
Implant stability | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway